CLINICAL TRIAL: NCT01646411
Title: Phase I Study for Positive IgM Antibody Detection in New Diagnostic Test Kit for for Acute Phase Infection
Brief Title: 300 Antibody Diagnostic Test Kit
Acronym: Antibody 300
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Plasma Source (Industry)
Collaborators: Plasma Services Group (Industry)
Responsible Party: Sponsor
Other Study IDs: 300831
Record Dates: First submitted 2012-07-12; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Acute Bacterial Infections; Acute Viral Infections
Keywords: cytomegalovirus (CMV) IgM &IgG; Lyme; Toxoplasma; Rubella; Rubeola IgM; Rocky mountain Spotted Fever IgM; Ebv IgM; Herpes; Babesia; Measles; Tetanus; Mumps; Mycoplasma; Legionella; Giardia; Syphilis; Bordetella Pertussis; H Pylori; Antibody Titre; Elevated IgG; Abnormal IgM; SLE
MeSH Terms: conditions — Hyper-IgM Immunodeficiency Syndrome, Type 1; Rubella; Herpes Simplex; Measles; Tetanus; Mumps; Mycoplasma Infections; Giardiasis; Syphilis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum collected in two 10ml sst and two 8ml edta venipuncture tubes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- assorted acute infection: 300 patients diagnosed with assorted acute infection.

SUMMARY:
For the development of a Point of Care IVD test kit for acute phase disease detection against a variety of bacterial and viral infections. Phase one includes 100 clinical diagnosed positive and 200 clinically "normal" serum and whole blood matched specimens for specificity and sensitivity determination for each marker. The positive samples must be IgM positive using any FDA cleared ELISA test kit. The negatives samples must be negative for IgM.

ELIGIBILITY:
Inclusion Criteria:

* current acute infection
* age 18-70
* male or female
* any race
* currently active symptoms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute infection between the age of 18 and 70. Sex and race are random.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
IgM greater than 1xcut off value | Antibody value measured within seven days of specimen collection.
  Elisa System positive results are greater than 1 times the cutoff. Negative less than 1x cutoff.
  Prevalence of IGM in general mid-atlantic population is less than 10% of study population.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Flieshman, M.S immunology, Study Director
Locations (1):
- The Plasma Source, Southampton, Pennsylvania, United States